CLINICAL TRIAL: NCT06668818
Title: Clinical Nursing Practice Supported by Results of Research: Mixed-method Study
Acronym: PRACTICE
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2023-83
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nurses employed at IRCCS-CRO Aviano
- Patients admitted to the IRCCS-CRO Aviano as in-patients

SUMMARY:
The purpose of the study is to assess the attitudes and the use of research by nurses at the IRCCS-CRO Aviano. Furthermore, it will make it possible to identify attitudes towards the use/non-use of research results, specific training needs and targeted interventions to ensure adequate care for cancer patients along the disease course, derived from a constant updating of nursing skills. The study will involve nurses working in different care settings of the Institute and some patients who will be able to express their care needs and research priorities, making a direct contribution towards development of care centred on the health needs, preferences and values of the cancer patients.

ELIGIBILITY:
Inclusion criteria for nurses:

* All nurses employed at IRCCS-CRO Aviano under fixed-term and permanent contract on 15 September 2023;
* Nursing activities in the departments of medical and surgical oncology and high technologies;
* Full-time and part-time employment contract;
* Signature of consent for participation in the study and processing of personal data (Privacy).

Patient inclusion criteria:

* Patients admitted to the institution as in-patients;
* Age ≥ 18 years;
* Signature of consent for participation in the study and processing of personal data (Privacy);
* Good understanding of the Italian language.

Exclusion criteria for nurses:

- Lack of willingness/interest in participating in the study and signing the consent.

Patient exclusion criteria:

* Day-Hospital patients;
* Age < 18 years;
* Diagnosis of cognitive dysfunction or psychiatric disorders;
* Difficulties in understanding the Italian language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurses employed at IRCCS-CRO Aviano and patients admitted to the institution as in-patients
Sampling Method: Non-Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2025-03-07 (Estimated); Study Completion 2025-03-07 (Estimated)

PRIMARY OUTCOMES:
To assess the attitudes and use of research by nurses IRCCS of Aviano | 1 year
  The Modified Research Utilization Questionnaire (M-RUQ), consisting of 22 items across three subscales assessed on a 5-point Likert scale (range: 22-110), will be used for data collection. Total scores are computed by summing and averaging domain scores, with reverse-scoring for negative items. Missing data will be imputed with item means, and results presented as mean ± standard deviation.

SECONDARY OUTCOMES:
To identify nursing issues, research priorities, and educational needs of nurses at IRCCS Aviano. | 1 year
  he qualitative data obtained from the research (using interview and focus group method) will be evaluated with inductive content analysis, following Colaizzi's framework (1978). In order to enhance the validity of the data, two researchers will independently examine the transcripts, and comprehensive readings will be conducted. Codes will be generated and compared by interpreting differences and similarities, from which themes and sub-themes will be obtained
To explore care needs and research priorities of patients at IRCCS Aviano | 1 year
  he qualitative data obtained from the research (using interview and focus group method) will be evaluated with inductive content analysis, following Colaizzi's framework (1978). In order to enhance the validity of the data, two researchers will independently examine the transcripts, and comprehensive readings will be conducted. Codes will be generated and compared by interpreting differences and similarities, from which themes and sub-themes will be obtained

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Cadorin, PhD, Principal Investigator — Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS
Locations (1):
- Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS, Aviano, Pordenone, Italy